CLINICAL TRIAL: NCT03735849
Title: A Phase 1 Clinical Trial to Evaluate the Safety and Pharmacokinetics of VRC-HIVMAB075-00-AB (VRC07-523LS) in the Sera and Mucosae of Healthy, HIV-1-Uninfected Adult Participants
Brief Title: Evaluating the Safety and Pharmacokinetics of VRC07-523LS in the Sera and Mucosae of Healthy, HIV-Uninfected Adult Participants
Acronym: VRC07-523LS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HVTN 128; 38523 (Registry Identifier: DAIDS-ES Registry Number)
Record Dates: First submitted 2018-11-07; First posted 2018-11-08 (Actual); Results first posted 2022-03-07 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Pre-treatment (No Intervention): Biopsy collected but was not randomized to any treatment group
- Group 1: VRC07-523LS (Experimental): Participants will receive 10 mg/kg of VRC07-523LS at Weeks 0, 16, and 32.
  Interventions: Biological: VRC07-523LS
- Group 2: VRC07-523LS (Experimental): Participants will receive 30 mg/kg of VRC07-523LS at Weeks 0, 16, and 32.
  Interventions: Biological: VRC07-523LS

INTERVENTIONS:
Biological: VRC07-523LS — Administered by intravenous (IV) infusion
  Other Names: VRC-HIVMAB075-00-AB
  Arms: Group 1: VRC07-523LS; Group 2: VRC07-523LS

SUMMARY:
The purpose of this study is to evaluate the safety and pharmacokinetics of a human monoclonal antibody (VRC07-523LS) in the sera and mucosae of healthy, HIV-uninfected adults.

DETAILED DESCRIPTION:
This study will evaluate the safety and pharmacokinetics of a human monoclonal antibody (VRC07-523LS) in the sera and mucosae of healthy, HIV-uninfected adults.

Participants will be randomly assigned to one of two groups. Participants in Group 1 will receive 10 mg/kg of VRC07-523LS at Weeks 0, 16, and 32. Participants in Group 2 will receive 30 mg/kg of VRC07-523LS at Weeks 0, 16, and 32.

Study visits will occur at Weeks 0, 2, 16, 18, 32, 34, and 48. Visits may include physical examinations; blood and urine collection; rectal, cervicovaginal, and seminal secretion collection; cervical, rectal, and vaginal biopsy collection; HIV testing; risk reduction counseling; and questionnaires. Study staff will contact participants at Week 50 for follow-up safety monitoring.

ELIGIBILITY:
Inclusion Criteria:

General and Demographic Criteria

* Age of 18 to 50 years
* Access to a participating HIV Vaccine Trials Network (HVTN) clinical research site (CRS) and willingness to be followed for the planned duration of the study
* Ability and willingness to provide informed consent
* Assessment of understanding: volunteer demonstrates understanding of this study and completes a questionnaire prior to first study product administration with verbal demonstration of understanding of all questionnaire items answered incorrectly
* Agrees not to enroll in another study of an investigational research agent until completion of the last required protocol clinic visit
* Good general health as shown by medical history, physical exam, and screening laboratory tests

HIV-Related Criteria:

* Willingness to receive HIV test results
* Willingness to discuss HIV infection risks and amenable to HIV risk reduction counseling.
* Assessed by the clinic staff as being at "low risk" for HIV infection and committed to maintaining behavior consistent with low risk of HIV exposure through the last required protocol clinic visit. See the study protocol for US Low risk guidelines.

Laboratory Inclusion Values

Hemogram/Complete blood count (CBC)

* Hemoglobin greater than or equal to 11.0 g/dL for volunteers who were assigned female sex at birth, greater than or equal to 13.0 g/dL for volunteers who were assigned male sex at birth. For transgender participants who have been on hormone therapy for more than 6 consecutive months, determine hemoglobin eligibility based on the gender with which they identify (ie, a transgender female who has been on feminizing hormone therapy for more than 6 consecutive months should be assessed for eligibility using the hemoglobin parameters for persons assigned female sex at birth).
* White blood cell (WBC) count equal to 2,500 to 12,000 cells/mm^3
* WBC differential either within institutional normal range or with site physician approval
* Platelets equal to 125,000 to 550,000/mm^3

Chemistry

* Chemistry panel: Alanine aminotransferase (ALT) less than 1.25 times the institutional upper limit of normal and creatinine less than or equal to institutional upper limits of normal.

Virology

* Negative HIV-1 and -2 blood test: US volunteers must have a negative US Food and Drug Administration (FDA)-approved enzyme immunoassay (EIA) or chemiluminescent microparticle immunoassay (CMIA).
* Negative Hepatitis B surface antigen (HBsAg)
* Negative anti-Hepatitis C virus (anti-HCV) antibodies, or negative HCV polymerase chain reaction (PCR) if the anti-HCV is positive

Urine

* Normal urine:

  * Negative or trace urine protein

Reproductive Status

* Volunteers who were assigned female sex at birth: negative serum or urine beta human chorionic gonadotropin (β-HCG) pregnancy test performed prior to biopsy collection and/or study product administration.
* Reproductive status: A volunteer who was assigned female sex at birth must:

  * Agree to use effective contraception for sexual activity that could lead to pregnancy from at least 21 days prior to enrollment through the last required protocol clinic visit. Effective contraception is defined as using the following methods:

    * Condoms (male or female) with or without a spermicide,
    * Diaphragm or cervical cap with spermicide,
    * Intrauterine device (IUD),
    * Hormonal contraception, or
    * Any other contraceptive method approved by the HVTN 128 Protocol Safety Review Team (PSRT)
    * Successful vasectomy in any partner assigned male sex at birth (considered successful if a volunteer reports that a male partner has [1] documentation of azoospermia by microscopy, or [2] a vasectomy more than 2 years ago with no resultant pregnancy despite sexual activity postvasectomy);
    * Tubal ligation
  * Or be sexually abstinent until at least 4 months following the last study product administration.
* Volunteers who were assigned female sex at birth must also agree not to seek pregnancy through alternative methods, such as artificial insemination or in vitro fertilization until after the last required protocol clinic visit

Mucosal Specimen Collection

* Volunteers 21 years of age and older who were assigned female sex at birth: Pap smear (verified by medical records) is required within:

  * the 3 years prior to enrollment with the latest result reported as normal or ASCUS (atypical squamous cells of undetermined significance), OR
  * the 5 years prior to enrollment, with the latest result reported as normal, or ASCUS with no evidence of high risk HPV.
* If no Pap smear was done within the last 3 years (or within the last 5 years, if high risk HPV testing was performed), the volunteer must be willing to undergo a Pap smear with the result reported (verified by medical records) as normal or ASCUS prior to sample collection.
* Willing to have mucosal secretions and tissue biopsies collected at several timepoints
* Willing to abstain from sexual intercourse for the required period after each biopsy collection

Exclusion Criteria:

General

* Weight greater than 115 kg
* Blood products received within 120 days before first study product administration unless eligibility for earlier enrollment is determined by the HVTN 128 PSRT
* Investigational research agents received within 30 days before first study product administration
* Intent to participate in another study of an investigational research agent or any other study that requires non-HVTN HIV antibody testing during the planned duration of the study
* Pregnant or breastfeeding

Vaccines and other Injections

* HIV vaccine(s) received in a prior HIV vaccine trial. For volunteers who have received control/placebo in an HIV vaccine trial, the HVTN 128 PSRT will determine eligibility on a case-by-case basis.
* Previous receipt of humanized or human monoclonal antibodies (mAbs), whether licensed or investigational; the HVTN 128 PSRT will determine eligibility on a case-by-case basis.
* Previous receipt of monoclonal antibodies against HIV

Immune System

* Immunosuppressive medications received within 30 days before first infusion (Not exclusionary: [1] corticosteroid nasal spray; [2] inhaled corticosteroids; [3] topical corticosteroids for mild, uncomplicated dermatitis; or [4] a single course of oral/parenteral prednisone or equivalent at doses less than or equal to 20 mg/day and length of therapy less than 14 days)
* Serious adverse reactions to VRC07-523LS formulation components (sucrose, histidine, and sorbitol; see study protocol for more information), including history of anaphylaxis and related symptoms such as hives, respiratory difficulty, angioedema, and/or abdominal pain.
* Immunoglobulin received within 90 days before first infusion unless eligibility for earlier enrollment is determined by the HVTN 128 PSRT
* Autoimmune disease (Not excluded from participation: Volunteer with mild, stable and uncomplicated autoimmune disease that does not require immunosuppressive medication and that, in the judgment of the site investigator, is likely not subject to exacerbation and likely not to complicate Solicited and Unsolicited AE assessments)
* Immunodeficiency

Clinically significant medical conditions

* Clinically significant medical condition, physical examination findings, clinically significant abnormal laboratory results, or past medical history with clinically significant implications for current health. A clinically significant condition or process includes but is not limited to:

  * A process that would affect the immune response,
  * A process that would require medication that affects the immune response,
  * Any contraindication to repeated infusions or blood draws, including inability to establish venous access,
  * A condition that requires active medical intervention or monitoring to avert grave danger to the volunteer's health or well-being during the study period,
  * A condition or process (eg, chronic urticaria or recent infusion with evidence of residual inflammation) for which signs or symptoms could be confused with reactions to the study product, or
  * Any condition specifically listed among the exclusion criteria below.
* Any medical, psychiatric, occupational, or other condition that, in the judgment of the investigator, would interfere with, or serve as a contraindication to, protocol adherence, assessment of safety, Solicited AEs, or a volunteer's ability to give informed consent
* Psychiatric condition that precludes compliance with the protocol. Specifically excluded are persons with psychoses within the past 3 years, ongoing risk for suicide, or history of suicide attempt or gesture within the past 3 years.
* Current anti-tuberculosis (TB) therapy
* Asthma other than mild, well-controlled asthma. (Symptoms of asthma severity as defined in the most recent National Asthma Education and Prevention Program (NAEPP) Expert Panel report). Exclude a volunteer who:

  * Uses a short-acting rescue inhaler (typically a beta 2 agonist) daily, or
  * Uses moderate/high dose inhaled corticosteroids, or
  * In the past year has either of the following:

    * Greater than 1 exacerbation of symptoms treated with oral/parenteral corticosteroids;
    * Needed emergency care, urgent care, hospitalization, or intubation for asthma.
* Diabetes mellitus type 1 or type 2. (Not excluded: type 2 cases controlled with diet alone or a history of isolated gestational diabetes.)
* Hypertension:

  * If a person has been found to have elevated blood pressure or hypertension during screening or previously, exclude for blood pressure that is not well controlled. Well-controlled blood pressure is defined as consistently less than or equal to 140 mm Hg systolic and less than or equal to 90 mm Hg diastolic, with or without medication, with only isolated, brief instances of higher readings, which must be less than or equal to 150 mm Hg systolic and less than or equal to 100 mm Hg diastolic. For these volunteers, blood pressure must be less than or equal to 140 mm Hg systolic and less than or equal to 90 mm Hg diastolic at enrollment.
  * If a person has NOT been found to have elevated blood pressure or hypertension during screening or previously, exclude for systolic blood pressure greater than or equal to 150 mm Hg at enrollment or diastolic blood pressure greater than or equal to 100 mm Hg at enrollment.
* Bleeding disorder diagnosed by a doctor (eg, factor deficiency, coagulopathy, or platelet disorder requiring special precautions)
* Malignancy (Not excluded from participation: Volunteer who has had malignancy excised surgically and who, in the investigator's estimation, has a reasonable assurance of sustained cure, or who is unlikely to experience recurrence of malignancy during the period of the study)
* Seizure disorder: History of seizure(s) within past three years. Also exclude if volunteer has used medications in order to prevent or treat seizure(s) at any time within the past 3 years
* Asplenia: any condition resulting in the absence of a functional spleen
* History of hereditary angioedema, acquired angioedema, or idiopathic angioedema.

Mucosal Specimen Collection

* A rectal condition (for rectal biopsies), such as an active infection or inflammation of the colorectal area (eg, an HSV-2 outbreak or inflamed hemorrhoids or colitis/diarrhea), internal hemorrhoids, or any other condition noted during screening rectal exam via anoscope or in medical history that in the opinion of the clinician represents a contraindication to mucosal sampling.
* For those who were assigned female sex at birth (for vaginal and cervical biopsies), any condition noted during pelvic exam via speculum or in medical history that in the opinion of the clinician represents a contraindication to mucosal sampling (eg, bacterial vaginosis).
* An active genital tract condition, such as an active infection or inflammation of the genital tract (eg, genital sores or ulcers, penile or abnormal vaginal discharge, genital warts that are symptomatic or requiring treatment) or any other condition that in the opinion of the clinician represents a contraindication to mucosal sampling.
* Hysterectomy or bilateral oophorectomy
* Menopause
* Current use of anticoagulants

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2019-01-18 (Actual); Primary Completion 2020-12-21 (Actual); Study Completion 2020-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Walsh, Study Chair — Brigham and Women's Hospital; Maria Lemos, Study Chair — Fred Hutch
Locations (2):
- United States (2):
  - Brigham and Women's Hospital Vaccine CRS (BWH VCRS), Boston, Massachusetts
  - Seattle Vaccine and Prevention CRS, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Vaccine: VRC07-523LS (VRC-HIVMAB075-00-AB) 10 mg/kg to be administered IV at weeks 0, 16, and 32
- Group 2: Vaccine: VRC07-523LS (VRC-HIVMAB075-00-AB) 30 mg/kg to be administered IV at weeks 0, 16, and 32
- Group 3: Pre-treatment: Biopsy collected but was not randomized to any treatment group
Period: Overall Study
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Pre-treatment
Started | 11 | 13 | 4
Safety Population | 11 | 13 | 4
Completed | 9 | 13 | 0
Not Completed | 2 | 0 | 4
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Participant unable to adhere to visit | 1 | 0 | 0
Not completed — Not Randomized | 0 | 0 | 4

BASELINE CHARACTERISTICS:
Population: Participants who have their biopsies collected
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Pre-treatment | Total
Number analyzed (Participants) | 11 | 13 | 4 | 28
Age, Continuous [Median (Full Range); unit: years] | 28 [23 to 45] | 26 [18 to 43] | 22 [18 to 30] | 26 [18 to 45]
Age, Customized [Count of Participants; unit: Participants]
  Less than 18 years | 0 | 0 | 0 | 0
  18 - 20 years | 0 | 3 | 2 | 5
  21 - 30 years | 6 | 6 | 2 | 14
  31 - 40 years | 4 | 1 | 0 | 5
  41 - 50 years | 1 | 3 | 0 | 4
  Above 50 years | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 1 | 13
  Male | 5 | 7 | 3 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 1 | 3
  Not Hispanic or Latino | 9 | 13 | 3 | 25
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 1 | 4
  White | 10 | 8 | 3 | 21
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  USA | 11 | 13 | 4 | 28

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Local Reactogenicity Signs and Symptoms
Description: Graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1, July 2017. The maximum grade observed for each symptom over the time frame is presented.
Time Frame: Measured through 3 days after each infusion at weeks 0, 16 and 32
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Vaccine | Group 2: Vaccine
Number analyzed (Participants) | 11 | 13
Participants
  Pain and/or Tenderness: None | 5 | 10
  Pain and/or Tenderness: Mild | 6 | 3
  Pain and/or Tenderness: Moderate | 0 | 0
  Pain and/or Tenderness: Severe | 0 | 0
  Pain and/or Tenderness: Potentially Life-threatening | 0 | 0
  Erythema: None | 10 | 12
  Erythema: Mild | 1 | 1
  Erythema: Moderate | 0 | 0
  Erythema: Severe | 0 | 0
  Erythema: Potentially Life-threatening | 0 | 0
  Induration: None | 11 | 12
  Induration: Mild | 0 | 1
  Induration: Moderate | 0 | 0
  Induration: Severe | 0 | 0
  Induration: Potentially Life-threatening | 0 | 0
  Erythema and/or Induration: None | 10 | 11
  Erythema and/or Induration: Mild | 1 | 2
  Erythema and/or Induration: Moderate | 0 | 0
  Erythema and/or Induration: Severe | 0 | 0
  Erythema and/or Induration: Potentially Life-threatening | 0 | 0

2. Primary Outcome: Number of Participants Reporting Systemic Reactogenicity Signs and Symptoms
Description: as for outcome 1
Time Frame: Measured through 3 days after each infusion at weeks 0, 16 and 32
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Vaccine | Group 2: Vaccine
Number analyzed (Participants) | 11 | 13
Participants
  Malaise and/or fatigue: None | 3 | 4
  Malaise and/or fatigue: Mild | 6 | 5
  Malaise and/or fatigue: Moderate | 2 | 3
  Malaise and/or fatigue: Severe | 0 | 1
  Malaise and/or fatigue: Potentially Life-threatening | 0 | 0
  Myalgia: None | 8 | 8
  Myalgia: Mild | 3 | 3
  Myalgia: Moderate | 0 | 1
  Myalgia: Severe | 0 | 1
  Myalgia: Potentially Life-threatening | 0 | 0
  Headache: None | 3 | 6
  Headache: Mild | 5 | 5
  Headache: Moderate | 3 | 2
  Headache: Severe | 0 | 0
  Headache: Potentially Life-threatening | 0 | 0
  Nausea: None | 6 | 10
  Nausea: Mild | 5 | 3
  Nausea: Moderate | 0 | 0
  Nausea: Severe | 0 | 0
  Nausea: Potentially Life-threatening | 0 | 0
  Chills: None | 9 | 7
  Chills: Mild | 1 | 3
  Chills: Moderate | 1 | 1
  Chills: Severe | 0 | 2
  Chills: Potentially Life-threatening | 0 | 0
  Arthralgia: None | 10 | 11
  Arthralgia: Mild | 1 | 1
  Arthralgia: Moderate | 0 | 0
  Arthralgia: Severe | 0 | 1
  Arthralgia: Potentially Life-threatening | 0 | 0
  Facial flushing: None | 8 | 12
  Facial flushing: Mild | 3 | 1
  Facial flushing: Moderate | 0 | 0
  Facial flushing: Severe | 0 | 0
  Facial flushing: Potentially Life-threatening | 0 | 0
  Non-exertional dyspnea: None | 11 | 12
  Non-exertional dyspnea: Mild | 0 | 1
  Non-exertional dyspnea: Moderate | 0 | 0
  Non-exertional dyspnea: Severe | 0 | 0
  Non-exertional dyspnea: Potentially Life-threatening | 0 | 0
  Urticaria: None | 11 | 13
  Urticaria: Mild | 0 | 0
  Urticaria: Moderate | 0 | 0
  Urticaria: Severe | 0 | 0
  Urticaria: Potentially Life-threatening | 0 | 0
  Non-exertional tachycardia: None | 10 | 13
  Non-exertional tachycardia: Mild | 1 | 0
  Non-exertional tachycardia: Moderate | 0 | 0
  Non-exertional tachycardia: Severe | 0 | 0
  Non-exertional tachycardia: Potentially Life-threatening | 0 | 0
  Generalized Pruritus: None | 11 | 12
  Generalized Pruritus: Mild | 0 | 0
  Generalized Pruritus: Moderate | 0 | 1
  Generalized Pruritus: Severe | 0 | 0
  Generalized Pruritus: Potentially Life-threatening | 0 | 0
  Unexplained diaphoresis: None | 10 | 13
  Unexplained diaphoresis: Mild | 1 | 0
  Unexplained diaphoresis: Moderate | 0 | 0
  Unexplained diaphoresis: Severe | 0 | 0
  Unexplained diaphoresis: Potentially Life-threatening | 0 | 0
  Max. Systemic Symptoms: None | 1 | 2
  Max. Systemic Symptoms: Mild | 5 | 7
  Max. Systemic Symptoms: Moderate | 5 | 2
  Max. Systemic Symptoms: Severe | 0 | 2
  Max. Systemic Symptoms: Potentially Life-threatening | 0 | 0
  Temperature: None | 10 | 11
  Temperature: Mild | 1 | 0
  Temperature: Moderate | 0 | 2
  Temperature: Severe | 0 | 0
  Temperature: Potentially Life-threatening | 0 | 0

3. Primary Outcome: Chemistry and Hematology Laboratory Measures - Alanine Aminotransferase (ALT) in U/L
Description: For each local laboratory measure, summary statistics were presented by treatment group and timepoint for the overall population.
Time Frame: Measured during screening, visit 4(day 14), 6 (day 126) and 8 (day 238)
Population: Samples were missing for follow-up visits due to miss visits or discontinuing study product.
Measure: Median (Inter-Quartile Range); unit: U/L
Arm/Group | Group 1: Vaccine | Group 2: Vaccine
Number analyzed (Participants) | 11 | 13
U/L
  ALT (SGPT) (U/L)- Screening | 19.0 [9.0 to 26.0] | 16.0 [11.0 to 20.0]
  ALT (SGPT) (U/L)-Day 14 | 14.0 [10.0 to 18.0] | 16.0 [12.0 to 24.0]
  ALT (SGPT) (U/L)-Day 126: number analyzed (Participants) | 10 | 13
  ALT (SGPT) (U/L)-Day 126 | 22.0 [13.0 to 24.0] | 17.0 [12.0 to 26.0]
  ALT (SGPT) (U/L)-Day 238: number analyzed (Participants) | 9 | 11
  ALT (SGPT) (U/L)-Day 238 | 16.0 [14.0 to 26.0] | 14.0 [11.0 to 23.0]

4. Primary Outcome: Chemistry and Hematology Laboratory Measures- Hemoglobin and Creatinine (g/dl)
Description: For each local laboratory measure-Hemoglobin and Creatinine (g/dl), summary statistics were presented by treatment group and time point for the overall population.
Time Frame: Measured during screening, Day 14, 126, 238
Population: Samples were missing for follow-up visits due to miss visits or discontinuing study product.
Measure: Median (Inter-Quartile Range); unit: g/dL
Arm/Group | Group 1: Vaccine | Group 2: Vaccine
Number analyzed (Participants) | 11 | 13
g/dL
  Hemoglobin (g/dL)- Screening | 14.3 [13.3 to 14.6] | 13.9 [12.9 to 15.0]
  Hemoglobin (g/dL)-Day 14 | 13.4 [13.2 to 14.9] | 13.2 [12.3 to 14.8]
  Hemoglobin (g/dL)-Day 126: number analyzed (Participants) | 10 | 13
  Hemoglobin (g/dL)-Day 126 | 13.9 [13.4 to 14.7] | 14.0 [12.4 to 15.0]
  Hemoglobin (g/dL)-Day 238: number analyzed (Participants) | 9 | 11
  Hemoglobin (g/dL)-Day 238 | 13.9 [13.6 to 14.3] | 13.2 [12.6 to 14.8]
  Creatinine (g/dL)- Screening | .00076 [.00071 to .00094] | .00078 [.00071 to .00093]
  Creatinine (g/dL)-Day 14 | .00082 [.00071 to .00091] | .00081 [.00076 to .00092]
  Creatinine (g/dL)-Day 126: number analyzed (Participants) | 10 | 13
  Creatinine (g/dL)-Day 126 | .00077 [.00070 to .00102] | .00081 [.00064 to .00095]
  Creatinine (g/dL)-Day 238: number analyzed (Participants) | 9 | 11
  Creatinine (g/dL)-Day 238 | .00070 [.00067 to .00084] | .00085 [.00067 to .00093]

5. Primary Outcome: Chemistry and Hematology Laboratory Measures- Lymphocyte Count, Neutrophil Count, Platelets, White Blood Cells (WBC)
Description: For each local laboratory measure lymphocyte count, neutrophil count, platelets, white blood cells (WBC) in 1000/ cubic mm summary statistics were presented by treatment group and time point
Time Frame: Measured during screening, Day 14, 126, 238
Population: Samples were missing for follow-up visits due to miss visits or discontinuing study product.
Measure: Median (Inter-Quartile Range); unit: 1000 cells/cubic mm
Arm/Group | Group 1: Vaccine | Group 2: Vaccine
Number analyzed (Participants) | 11 | 13
1000 cells/cubic mm
  WBC (1000 cells/cubic mm)- Screening | 8.03 [5.91 to 8.77] | 7.12 [5.43 to 7.41]
  WBC (1000 cells/cubic mm)-Day 14 | 6.22 [5.18 to 8.77] | 7.12 [5.65 to 7.50]
  WBC (1000 cells/cubic mm)-Day 126: number analyzed (Participants) | 10 | 13
  WBC (1000 cells/cubic mm)-Day 126 | 7.63 [6.35 to 8.46] | 5.55 [5.35 to 6.21]
  WBC (1000 cells/cubic mm)-Day 238: number analyzed (Participants) | 9 | 11
  WBC (1000 cells/cubic mm)-Day 238 | 8.02 [6.88 to 8.42] | 5.22 [4.54 to 5.94]
  Neutrophils (1000 cells/cubic mm)- Screening | 4.74 [3.11 to 5.53] | 3.45 [3.00 to 4.89]
  Neutrophils (1000 cells/cubic mm)-Day 14 | 3.65 [3.25 to 5.85] | 3.90 [3.17 to 4.82]
  Neutrophils (1000 cells/cubic mm)-Day 126: number analyzed (Participants) | 10 | 13
  Neutrophils (1000 cells/cubic mm)-Day 126 | 4.98 [4.20 to 5.45] | 3.19 [2.99 to 3.72]
  Neutrophils (1000 cells/cubic mm)-Day 238: number analyzed (Participants) | 9 | 11
  Neutrophils (1000 cells/cubic mm)-Day 238 | 4.75 [3.92 to 6.29] | 3.10 [1.99 to 3.43]
  Lymphocytes (1000 cells/cubic mm)- Screening | 2.30 [1.39 to 2.45] | 2.28 [1.63 to 2.67]
  Lymphocytes (1000 cells/cubic mm)-Day 14 | 1.91 [1.20 to 2.51] | 1.82 [1.73 to 2.31]
  Lymphocytes (1000 cells/cubic mm)-Day 126: number analyzed (Participants) | 10 | 13
  Lymphocytes (1000 cells/cubic mm)-Day 126 | 1.72 [1.41 to 2.37] | 1.71 [1.18 to 2.19]
  Lymphocytes (1000 cells/cubic mm)-Day 238: number analyzed (Participants) | 9 | 11
  Lymphocytes (1000 cells/cubic mm)-Day 238 | 2.04 [1.50 to 2.27] | 1.64 [1.14 to 2.02]
  Platelets (1000 cells/cubic mm)- Screening | 260 [224 to 293] | 249 [215 to 273]
  Platelets (1000 cells/cubic mm)-Day 14 | 243 [215 to 291] | 225 [213 to 279]
  Platelets (1000 cells/cubic mm)-Day 126: number analyzed (Participants) | 10 | 13
  Platelets (1000 cells/cubic mm)-Day 126 | 247 [226 to 263] | 253 [221 to 280]
  Platelets (1000 cells/cubic mm)-Day 238: number analyzed (Participants) | 9 | 11
  Platelets (1000 cells/cubic mm)-Day 238 | 239 [230 to 271] | 264 [206 to 300]

6. Primary Outcome: Chemistry and Hematology Laboratory Measures
Description: Counts of lab grade >1 for ALT, creatine, hemoglobin, lymphocyte count, neutrophil, platelets, white blood cells
Time Frame: Measured during screening, Day 14, 126, 238
Population: Samples were missing for follow-up visits due to miss visits or discontinuing study product.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Vaccine | Group 2: Vaccine
Number analyzed (Participants) | 11 | 13
Participants
  WBC (1000 cells/cubic mm)- Screening | 0 | 0
  WBC (1000 cells/cubic mm)-Day 14 | 0 | 0
  WBC (1000 cells/cubic mm)-Day 126: number analyzed (Participants) | 10 | 13
  WBC (1000 cells/cubic mm)-Day 126 | 0 | 0
  WBC (1000 cells/cubic mm)-Day 238: number analyzed (Participants) | 9 | 11
  WBC (1000 cells/cubic mm)-Day 238 | 0 | 0
  Neutrophils (1000 cells/cubic mm)- Screening | 0 | 0
  Neutrophils (1000 cells/cubic mm)-Day 14 | 0 | 0
  Neutrophils (1000 cells/cubic mm)-Day 126: number analyzed (Participants) | 10 | 13
  Neutrophils (1000 cells/cubic mm)-Day 126 | 0 | 0
  Neutrophils (1000 cells/cubic mm)-Day 238: number analyzed (Participants) | 9 | 11
  Neutrophils (1000 cells/cubic mm)-Day 238 | 0 | 0
  Hemoglobin (g/dL)- Screening | 0 | 0
  Hemoglobin (g/dL)-Day 14 | 0 | 0
  Hemoglobin (g/dL)-Day 126: number analyzed (Participants) | 10 | 13
  Hemoglobin (g/dL)-Day 126 | 0 | 0
  Hemoglobin (g/dL)-Day 238: number analyzed (Participants) | 9 | 11
  Hemoglobin (g/dL)-Day 238 | 0 | 0
  Lymphocytes (1000 cells/cubic mm)- Screening | 0 | 0
  Lymphocytes (1000 cells/cubic mm)-Day 14 | 0 | 0
  Lymphocytes (1000 cells/cubic mm)-Day 126: number analyzed (Participants) | 10 | 13
  Lymphocytes (1000 cells/cubic mm)-Day 126 | 0 | 0
  Lymphocytes (1000 cells/cubic mm)-Day 238: number analyzed (Participants) | 9 | 11
  Lymphocytes (1000 cells/cubic mm)-Day 238 | 0 | 0
  Platelets (1000 cells/cubic mm)- Screening | 0 | 0
  Platelets (1000 cells/cubic mm)-Day 14 | 0 | 0
  Platelets (1000 cells/cubic mm)-Day 126: number analyzed (Participants) | 10 | 13
  Platelets (1000 cells/cubic mm)-Day 126 | 0 | 0
  Platelets (1000 cells/cubic mm)-Day 238: number analyzed (Participants) | 9 | 11
  Platelets (1000 cells/cubic mm)-Day 238 | 0 | 0
  ALT (SGPT) (U/L)- Screening | 0 | 0
  ALT (SGPT) (U/L)-Day 14 | 0 | 0
  ALT (SGPT) (U/L)-Day 126: number analyzed (Participants) | 10 | 13
  ALT (SGPT) (U/L)-Day 126 | 0 | 0
  ALT (SGPT) (U/L)-Day 238: number analyzed (Participants) | 9 | 11
  ALT (SGPT) (U/L)-Day 238 | 0 | 0
  Creatinine (g/dL)- Screening | 0 | 0
  Creatinine (g/dL)-Day 14 | 0 | 0
  Creatinine (g/dL)-Day 126: number analyzed (Participants) | 10 | 13
  Creatinine (g/dL)-Day 126 | 1 | 0
  Creatinine (g/dL)-Day 238: number analyzed (Participants) | 9 | 11
  Creatinine (g/dL)-Day 238 | 0 | 0

7. Primary Outcome: Number of Participants Reporting Adverse Events (AEs)
Description: Participants Max severity reported per participant over visit.
Time Frame: Enrollment through week 48
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Vaccine | Group 2: Vaccine
Number analyzed (Participants) | 11 | 13
Participants
  Mild | 1 | 4
  Moderate | 9 | 6
  Severe | 0 | 2
  Potentially life-threatening | 0 | 0
  No AE reported | 1 | 1

8. Primary Outcome: Number of Participants With Early Discontinuation of Vaccinations and Reason for Discontinuation
Description: The number (percentage) of participants with early discontinuation of vaccinations and reason for discontinuation was summarized by arm
Time Frame: Enrollment through last scheduled dose at week 32
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Vaccine | Group 2: Vaccine
Number analyzed (Participants) | 11 | 13
Participants
  Clinical event (not reacto, HIV, death) | 0 | 2
  Subject unable to attend clinic visits | 1 | 0
  Did not discontinue SPA | 10 | 11

9. Primary Outcome: Unnormalized Levels of VRC07-523LS in Genital and Rectal Secretions, as Well as Cervical, Vaginal, and Rectal Tissues at the Collection Timepoints
Description: Pharmacokinetic - Single Molecule Counting (PK-SMC) assay were used to measure passively infused VRC07-523LS broadly neutralizing monoclonal antibody in participant mucosa (secretions and biopsies) using 5C9 anti-idiotype antibody (anti-ID). Outcome measure is the concentration of VRC07-523LS.
Time Frame: Measured at Visits 2, 4, 5, 6, 7, 8, 9 (Weeks -2, 2, 16, 18, 32, 34, 48) in secretion samples (semen, cervicovaginal, and rectal) and at Visits 2, 4, 8, 9 (Weeks -2, 2, 34, 48) in biopsy samples (rectal, cervical, and vaginal).
Population: Overall Number of Participants Analyzed represents the total number of infused participants in each group. Within each group, data are presented separately by sex, so the Number Analyzed per Row reflects the number of participants within each sex subgroup who contributed data for a specific timepoint or measure. Subgroup counts may be smaller than the overall number due to this stratification and the application of assay-specific quality control criteria at each timepoint.
Measure: Median (Inter-Quartile Range); unit: µg/mL
Arm/Group | Group 1: Vaccine | Group 2: Vaccine
Number analyzed (Participants) | 11 | 13
µg/mL
  Cervical Biopsy-Female-Visit 2: number analyzed (Participants) | 6 | 6
  Cervical Biopsy-Female-Visit 2 | 1153.16 [1153.16 to 1153.16] | 1153.16 [1153.16 to 1153.16]
  Cervical Biopsy-Female-Visit 4: number analyzed (Participants) | 6 | 4
  Cervical Biopsy-Female-Visit 4 | 70184.27 [35745.15 to 126879.8] | 178305 [121589.3 to 401886.0]
  Cervical Biopsy-Female-Visit 8: number analyzed (Participants) | 6 | 5
  Cervical Biopsy-Female-Visit 8 | 57049.38 [46153.70 to 166880.5] | 175382.4 [102097.3 to 322539.0]
  Cervical Biopsy-Female-Visit 9: number analyzed (Participants) | 5 | 4
  Cervical Biopsy-Female-Visit 9 | 32941.43 [1153.16 to 45682.22] | 53680.14 [22712.45 to 83060.03]
  Rectal Biopsy-Female-Visit 2: number analyzed (Participants) | 6 | 6
  Rectal Biopsy-Female-Visit 2 | 1153.16 [1153.16 to 1153.16] | 1153.16 [1153.16 to 1153.16]
  Rectal Biopsy-Female-Visit 4: number analyzed (Participants) | 6 | 6
  Rectal Biopsy-Female-Visit 4 | 202976.8 [177021.1 to 210773.2] | 568748 [543576.9 to 623879.0]
  Rectal Biopsy-Female-Visit 8: number analyzed (Participants) | 6 | 5
  Rectal Biopsy-Female-Visit 8 | 182851.1 [151294.8 to 235197.4] | 715593.4 [470775.6 to 736740.7]
  Rectal Biopsy-Female-Visit 9: number analyzed (Participants) | 6 | 4
  Rectal Biopsy-Female-Visit 9 | 18611.77 [1153.16 to 36971.61] | 80218.02 [64065.28 to 94174.95]
  Rectal Biopsy-Male-Visit 2: number analyzed (Participants) | 5 | 6
  Rectal Biopsy-Male-Visit 2 | 1153.16 [1153.16 to 1153.16] | 1153.16 [1153.16 to 1153.16]
  Rectal Biopsy-Male-Visit 4: number analyzed (Participants) | 5 | 7
  Rectal Biopsy-Male-Visit 4 | 134874.1 [42174.80 to 219166.6] | 219156.5 [168027.4 to 430497.1]
  Rectal Biopsy-Male-Visit 8: number analyzed (Participants) | 3 | 5
  Rectal Biopsy-Male-Visit 8 | 284185.5 [195676.0 to 319445.8] | 641581.4 [556010.9 to 683383.9]
  Rectal Biopsy-Male-Visit 9: number analyzed (Participants) | 4 | 6
  Rectal Biopsy-Male-Visit 9 | 34940.14 [20126.11 to 43457.49] | 56888.7 [36844.67 to 95985.49]
  Rectal Secretions-Female-Visit 2: number analyzed (Participants) | 5 | 4
  Rectal Secretions-Female-Visit 2 | 1153.16 [1153.16 to 1153.16] | 1153.16 [1153.16 to 1153.16]
  Rectal Secretions-Female-Visit 4: number analyzed (Participants) | 6 | 4
  Rectal Secretions-Female-Visit 4 | 1153.16 [1153.16 to 1153.16] | 1153.16 [1153.16 to 1153.16]
  Rectal Secretions-Female-Visit 5: number analyzed (Participants) | 3 | 4
  Rectal Secretions-Female-Visit 5 | 1153.16 [1153.16 to 1153.16] | 1153.16 [1153.16 to 1153.16]
  Rectal Secretions-Female-Visit 6: number analyzed (Participants) | 3 | 4
  Rectal Secretions-Female-Visit 6 | 1153.16 [1153.16 to 1153.16] | 1153.16 [1153.16 to 1153.16]
  Rectal Secretions-Female-Visit 7: number analyzed (Participants) | 3 | 4
  Rectal Secretions-Female-Visit 7 | 1153.16 [1153.16 to 1153.16] | 1153.16 [1153.16 to 1153.16]
  Rectal Secretions-Female-Visit 8: number analyzed (Participants) | 5 | 6
  Rectal Secretions-Female-Visit 8 | 1153.16 [1153.16 to 1153.16] | 1153.16 [1153.16 to 1153.16]
  Rectal Secretions-Female-Visit 9: number analyzed (Participants) | 6 | 4
  Rectal Secretions-Female-Visit 9 | 1153.16 [1153.16 to 1153.16] | 1153.16 [1153.16 to 1153.16]
  Rectal Secretions-Male-Visit 2: number analyzed (Participants) | 4 | 6
  Rectal Secretions-Male-Visit 2 | 1153.16 [1153.16 to 1153.16] | 1153.16 [1153.16 to 1153.16]
  Rectal Secretions-Male-Visit 4: number analyzed (Participants) | 3 | 7
  Rectal Secretions-Male-Visit 4 | 1153.16 [1153.16 to 1153.16] | 1153.16 [1153.16 to 1153.16]
  Rectal Secretions-Male-Visit 5: number analyzed (Participants) | 3 | 6
  Rectal Secretions-Male-Visit 5 | 1153.16 [1153.16 to 1153.16] | 1153.16 [1153.16 to 1153.16]
  Rectal Secretions-Male-Visit 6: number analyzed (Participants) | 2 | 6
  Rectal Secretions-Male-Visit 6 | 1153.16 [1153.16 to 1153.16] | 1153.16 [1153.16 to 1153.16]
  Rectal Secretions-Male-Visit 7: number analyzed (Participants) | 3 | 5
  Rectal Secretions-Male-Visit 7 | 1153.16 [1153.16 to 1153.16] | 1153.16 [1153.16 to 1153.16]
  Rectal Secretions-Male-Visit 8: number analyzed (Participants) | 1 | 2
  Rectal Secretions-Male-Visit 8 | 1153.16 [1153.16 to 1153.16] | 1153.16 [1153.16 to 1153.16]
  Rectal Secretions-Male-Visit 9: number analyzed (Participants) | 2 | 5
  Rectal Secretions-Male-Visit 9 | 1153.16 [1153.16 to 1153.16] | 1153.16 [1153.16 to 1153.16]
  Semen-Male-Visit 2: number analyzed (Participants) | 5 | 7
  Semen-Male-Visit 2 | 461.26 [461.26 to 461.26] | 461.26 [461.26 to 461.26]
  Semen-Male-Visit 4: number analyzed (Participants) | 5 | 7
  Semen-Male-Visit 4 | 214747.1 [199223.5 to 227049.4] | 329345.7 [249175.5 to 625128.3]
  Semen-Male-Visit 5: number analyzed (Participants) | 4 | 6
  Semen-Male-Visit 5 | 34446.39 [30663.42 to 55936.20] | 81633.99 [55119.07 to 123155.9]
  Semen-Male-Visit 6: number analyzed (Participants) | 4 | 6
  Semen-Male-Visit 6 | 317137.1 [269689.4 to 365345.4] | 579910.8 [519728.2 to 660392.1]
  Semen-Male-Visit 7: number analyzed (Participants) | 4 | 6
  Semen-Male-Visit 7 | 48960.51 [37631.99 to 60626.10] | 70942.9 [48683.17 to 99838.85]
  Semen-Male-Visit 8: number analyzed (Participants) | 3 | 5
  Semen-Male-Visit 8 | 265248.3 [205725.2 to 291173.4] | 518469.9 [344545.0 to 610333.2]
  Semen-Male-Visit 9: number analyzed (Participants) | 4 | 6
  Semen-Male-Visit 9 | 60255.85 [47412.77 to 79063.26] | 87682.25 [38238.46 to 185159.1]
  Softcup Fluid-Female-Visit 2: number analyzed (Participants) | 4 | 5
  Softcup Fluid-Female-Visit 2 | 1153.16 [1153.16 to 26506.86] | 1153.16 [1153.16 to 38269.62]
  Softcup Fluid-Female-Visit 4: number analyzed (Participants) | 5 | 5
  Softcup Fluid-Female-Visit 4 | 1310855 [861547.6 to 2562996] | 5006078 [2617554 to 44842195]
  Softcup Fluid-Female-Visit 5: number analyzed (Participants) | 5 | 3
  Softcup Fluid-Female-Visit 5 | 201939.7 [187546.5 to 244570.1] | 436561.2 [352180.6 to 518304.3]
  Softcup Fluid-Female-Visit 6: number analyzed (Participants) | 5 | 6
  Softcup Fluid-Female-Visit 6 | 4357902 [3453944 to 5201059] | 2999531 [2534151 to 7238536]
  Softcup Fluid-Female-Visit 7: number analyzed (Participants) | 5 | 4
  Softcup Fluid-Female-Visit 7 | 1025192 [751975.2 to 1102886] | 649319.1 [279858.1 to 5294497]
  Softcup Fluid-Female-Visit 8: number analyzed (Participants) | 5 | 6
  Softcup Fluid-Female-Visit 8 | 2861361 [2774501 to 5461087] | 2640954 [2132056 to 3999627]
  Softcup Fluid-Female-Visit 9: number analyzed (Participants) | 2 | 3
  Softcup Fluid-Female-Visit 9 | 531608.8 [280123.4 to 783094.2] | 176998.6 [153141.8 to 597229.0]
  Vaginal Biopsy-Female-Visit 2: number analyzed (Participants) | 6 | 6
  Vaginal Biopsy-Female-Visit 2 | 1153.16 [1153.16 to 1153.16] | 1153.16 [1153.16 to 1153.16]
  Vaginal Biopsy-Female-Visit 4: number analyzed (Participants) | 6 | 4
  Vaginal Biopsy-Female-Visit 4 | 130086.2 [81265.22 to 147405.1] | 247847.2 [184451.4 to 363720.2]
  Vaginal Biopsy-Female-Visit 8: number analyzed (Participants) | 6 | 5
  Vaginal Biopsy-Female-Visit 8 | 105012 [52614.97 to 146829.3] | 111503.2 [1153.16 to 130445.6]
  Vaginal Biopsy-Female-Visit 9: number analyzed (Participants) | 5 | 4
  Vaginal Biopsy-Female-Visit 9 | 30650.35 [1153.16 to 44028.03] | 24562.42 [1153.16 to 48930.89]

10. Primary Outcome: IgG-normalized Levels of VRC07-523LS in Genital and Rectal Secretions, as Well as Cervical, Vaginal, and Rectal Tissues at the Collection Timepoints
Description: Pharmacokinetic - Single Molecule Counting (PK-SMC) assay were used to measure passively infused VRC07-523LS broadly neutralizing monoclonal antibody in participant mucosa (secretions and biopsies) using 5C9 anti-idiotype antibody (anti-ID). Outcome measure is the IgG-normalized VRC07-523LS levels performed by dividing VRC07-523LS levels (pg/mL) by the total IgG (ng/mL).
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: pg mAb/ng total IgG
Arm/Group | Group 1: Vaccine | Group 2: Vaccine
Number analyzed (Participants) | 11 | 13
pg mAb/ng total IgG
  Cervical Biopsy-Female-Visit 2: number analyzed (Participants) | 6 | 6
  Cervical Biopsy-Female-Visit 2 | 0.062 [0.039 to 0.1] | 0.047 [0.021 to 0.08]
  Cervical Biopsy-Female-Visit 4: number analyzed (Participants) | 6 | 4
  Cervical Biopsy-Female-Visit 4 | 3.92 [2.81 to 4.46] | 8.28 [7.56 to 10.33]
  Cervical Biopsy-Female-Visit 8: number analyzed (Participants) | 6 | 5
  Cervical Biopsy-Female-Visit 8 | 5.52 [4.62 to 6.29] | 11.56 [7.8 to 13.53]
  Cervical Biopsy-Female-Visit 9: number analyzed (Participants) | 5 | 4
  Cervical Biopsy-Female-Visit 9 | 0.84 [0.56 to 1.2] | 2.18 [1.58 to 2.42]
  Rectal Biopsy-Female-Visit 2: number analyzed (Participants) | 6 | 6
  Rectal Biopsy-Female-Visit 2 | 0.085 [0.075 to 0.11] | 0.09 [0.071 to 0.095]
  Rectal Biopsy-Female-Visit 4: number analyzed (Participants) | 6 | 6
  Rectal Biopsy-Female-Visit 4 | 9.8 [7.95 to 12.25] | 37.18 [30.12 to 41.68]
  Rectal Biopsy-Female-Visit 8: number analyzed (Participants) | 6 | 5
  Rectal Biopsy-Female-Visit 8 | 12.41 [10.2 to 13.97] | 44.02 [34.79 to 47.84]
  Rectal Biopsy-Female-Visit 9: number analyzed (Participants) | 6 | 4
  Rectal Biopsy-Female-Visit 9 | 1.02 [0.13 to 2.22] | 5.46 [5.19 to 5.78]
  Rectal Biopsy-Male-Visit 2: number analyzed (Participants) | 5 | 6
  Rectal Biopsy-Male-Visit 2 | 0.05 [0.048 to 0.057] | 0.07 [0.056 to 0.082]
  Rectal Biopsy-Male-Visit 4: number analyzed (Participants) | 5 | 7
  Rectal Biopsy-Male-Visit 4 | 8.35 [7.33 to 10.18] | 23.4 [18.91 to 27.21]
  Rectal Biopsy-Male-Visit 8: number analyzed (Participants) | 3 | 5
  Rectal Biopsy-Male-Visit 8 | 16.05 [13.81 to 16.45] | 41.92 [35.04 to 45.7]
  Rectal Biopsy-Male-Visit 9: number analyzed (Participants) | 4 | 6
  Rectal Biopsy-Male-Visit 9 | 2.34 [1.74 to 2.4] | 4.22 [1.54 to 7.49]
  Rectal Secretions-Female-Visit 2: number analyzed (Participants) | 5 | 4
  Rectal Secretions-Female-Visit 2 | 1.1 [0.93 to 1.76] | 4.39 [0.91 to 10.43]
  Rectal Secretions-Female-Visit 4: number analyzed (Participants) | 6 | 4
  Rectal Secretions-Female-Visit 4 | 0.96 [0.75 to 1.86] | 7.05 [2.24 to 11.44]
  Rectal Secretions-Female-Visit 5: number analyzed (Participants) | 3 | 4
  Rectal Secretions-Female-Visit 5 | 2.26 [1.6 to 7.7] | 3.22 [2.46 to 7.5]
  Rectal Secretions-Female-Visit 6: number analyzed (Participants) | 3 | 4
  Rectal Secretions-Female-Visit 6 | 1.43 [1.3 to 1.51] | 4.08 [1.87 to 6.09]
  Rectal Secretions-Female-Visit 7: number analyzed (Participants) | 3 | 4
  Rectal Secretions-Female-Visit 7 | 2.22 [1.44 to 6.83] | 2.77 [1.79 to 5.48]
  Rectal Secretions-Female-Visit 8: number analyzed (Participants) | 5 | 6
  Rectal Secretions-Female-Visit 8 | 2.79 [2.23 to 3.44] | 2.01 [1.62 to 4.23]
  Rectal Secretions-Female-Visit 9: number analyzed (Participants) | 6 | 4
  Rectal Secretions-Female-Visit 9 | 1.89 [1.19 to 2.65] | 1.51 [0.99 to 4.09]
  Rectal Secretions-Male-Visit 2: number analyzed (Participants) | 4 | 6
  Rectal Secretions-Male-Visit 2 | 1.86 [1.41 to 2.84] | 0.66 [0.35 to 0.72]
  Rectal Secretions-Male-Visit 4: number analyzed (Participants) | 3 | 7
  Rectal Secretions-Male-Visit 4 | 4.29 [3 to 5.15] | 0.92 [0.72 to 1.28]
  Rectal Secretions-Male-Visit 5: number analyzed (Participants) | 3 | 6
  Rectal Secretions-Male-Visit 5 | 4.43 [3.77 to 6.17] | 1.07 [0.85 to 2.88]
  Rectal Secretions-Male-Visit 6: number analyzed (Participants) | 2 | 6
  Rectal Secretions-Male-Visit 6 | 3.62 [2.45 to 4.79] | 2.38 [1.92 to 3.23]
  Rectal Secretions-Male-Visit 7: number analyzed (Participants) | 3 | 5
  Rectal Secretions-Male-Visit 7 | 5.8 [3.04 to 8.14] | 0.63 [0.43 to 1.86]
  Rectal Secretions-Male-Visit 8: number analyzed (Participants) | 1 | 2
  Rectal Secretions-Male-Visit 8 | 0.6 [0.6 to 0.6] | 2.56 [1.78 to 3.35]
  Rectal Secretions-Male-Visit 9: number analyzed (Participants) | 2 | 5
  Rectal Secretions-Male-Visit 9 | 2.18 [2.12 to 2.25] | 2.58 [0.89 to 3.78]
  Semen-Male-Visit 2: number analyzed (Participants) | 5 | 7
  Semen-Male-Visit 2 | 0.022 [0.017 to 0.027] | 0.03 [0.025 to 0.039]
  Semen-Male-Visit 4: number analyzed (Participants) | 5 | 7
  Semen-Male-Visit 4 | 9.08 [5.24 to 10.88] | 27.43 [14.99 to 28.27]
  Semen-Male-Visit 5: number analyzed (Participants) | 4 | 6
  Semen-Male-Visit 5 | 1.62 [1.53 to 2.34] | 3.57 [2.73 to 4.97]
  Semen-Male-Visit 6: number analyzed (Participants) | 4 | 6
  Semen-Male-Visit 6 | 16.09 [11.75 to 19.11] | 26.85 [22.29 to 33.2]
  Semen-Male-Visit 7: number analyzed (Participants) | 4 | 6
  Semen-Male-Visit 7 | 2.44 [1.86 to 3.42] | 2.71 [2.09 to 5.7]
  Semen-Male-Visit 8: number analyzed (Participants) | 3 | 5
  Semen-Male-Visit 8 | 14.07 [11.04 to 15.81] | 28.18 [25.16 to 33.77]
  Semen-Male-Visit 9: number analyzed (Participants) | 4 | 6
  Semen-Male-Visit 9 | 2.76 [2.26 to 3.23] | 2.95 [1.74 to 6.46]
  Softcup Fluid-Female-Visit 2: number analyzed (Participants) | 4 | 5
  Softcup Fluid-Female-Visit 2 | 0.0068 [0.0054 to 0.028] | 0.009 [0.0018 to 0.079]
  Softcup Fluid-Female-Visit 4: number analyzed (Participants) | 5 | 5
  Softcup Fluid-Female-Visit 4 | 3.74 [2.77 to 6.82] | 14.74 [12.99 to 21.47]
  Softcup Fluid-Female-Visit 5: number analyzed (Participants) | 5 | 3
  Softcup Fluid-Female-Visit 5 | 0.71 [0.67 to 0.75] | 2.75 [1.83 to 2.81]
  Softcup Fluid-Female-Visit 6: number analyzed (Participants) | 5 | 6
  Softcup Fluid-Female-Visit 6 | 6.8 [6.41 to 9.1] | 15.66 [11.02 to 18.49]
  Softcup Fluid-Female-Visit 7: number analyzed (Participants) | 5 | 4
  Softcup Fluid-Female-Visit 7 | 1.6 [0.88 to 2.65] | 1.73 [0.81 to 4.34]
  Softcup Fluid-Female-Visit 8: number analyzed (Participants) | 5 | 6
  Softcup Fluid-Female-Visit 8 | 7.15 [4.64 to 8.69] | 18.05 [12.38 to 20.9]
  Softcup Fluid-Female-Visit 9: number analyzed (Participants) | 2 | 3
  Softcup Fluid-Female-Visit 9 | 0.88 [0.54 to 1.21] | 1.38 [1 to 2.18]
  Vaginal Biopsy-Female-Visit 2: number analyzed (Participants) | 6 | 6
  Vaginal Biopsy-Female-Visit 2 | 0.059 [0.044 to 0.098] | 0.23 [0.073 to 0.48]
  Vaginal Biopsy-Female-Visit 4: number analyzed (Participants) | 6 | 4
  Vaginal Biopsy-Female-Visit 4 | 4.85 [4.61 to 5.67] | 14.49 [11.25 to 14.66]
  Vaginal Biopsy-Female-Visit 8: number analyzed (Participants) | 6 | 5
  Vaginal Biopsy-Female-Visit 8 | 7.41 [5.85 to 8.53] | 11.41 [0.83 to 16.54]
  Vaginal Biopsy-Female-Visit 9: number analyzed (Participants) | 5 | 4
  Vaginal Biopsy-Female-Visit 9 | 1.29 [0.33 to 1.49] | 3.01 [2.53 to 4.81]

11. Primary Outcome: Protein-normalized Levels of VRC07-523LS in Genital and Rectal Secretions, as Well as Cervical, Vaginal, and Rectal Tissues at the Collection Timepoints
Description: Pharmacokinetic - Single Molecule Counting (PK-SMC) assay were used to measure passively infused VRC07-523LS broadly neutralizing monoclonal antibody in participant mucosa (secretions and biopsies) using 5C9 anti-idiotype antibody (anti-ID). Outcome measure is the protein-normalized VRC07-523LS levels performed by dividing VRC07-523LS levels (pg/mL) by the total protein (ng/mL).
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: pg mAb/ng total protein
Arm/Group | Group 1: Vaccine | Group 2: Vaccine
Number analyzed (Participants) | 11 | 13
pg mAb/ng total protein
  Cervical Biopsy-Female-Visit 2: number analyzed (Participants) | 6 | 6
  Cervical Biopsy-Female-Visit 2 | 0.0024 [0.0018 to 0.0033] | 0.0018 [0.001 to 0.0029]
  Cervical Biopsy-Female-Visit 4: number analyzed (Participants) | 6 | 4
  Cervical Biopsy-Female-Visit 4 | 0.12 [0.086 to 0.18] | 0.32 [0.27 to 0.49]
  Cervical Biopsy-Female-Visit 8: number analyzed (Participants) | 6 | 5
  Cervical Biopsy-Female-Visit 8 | 0.16 [0.12 to 0.24] | 0.36 [0.3 to 0.5]
  Cervical Biopsy-Female-Visit 9: number analyzed (Participants) | 5 | 4
  Cervical Biopsy-Female-Visit 9 | 0.054 [0.0051 to 0.056] | 0.086 [0.052 to 0.12]
  Rectal Biopsy-Female-Visit 2: number analyzed (Participants) | 6 | 6
  Rectal Biopsy-Female-Visit 2 | 0.0014 [0.0012 to 0.0014] | 0.0011 [0.001 to 0.0012]
  Rectal Biopsy-Female-Visit 4: number analyzed (Participants) | 6 | 6
  Rectal Biopsy-Female-Visit 4 | 0.14 [0.14 to 0.15] | 0.49 [0.46 to 0.51]
  Rectal Biopsy-Female-Visit 8: number analyzed (Participants) | 6 | 5
  Rectal Biopsy-Female-Visit 8 | 0.17 [0.16 to 0.19] | 0.58 [0.46 to 0.62]
  Rectal Biopsy-Female-Visit 9: number analyzed (Participants) | 6 | 4
  Rectal Biopsy-Female-Visit 9 | 0.014 [0.0019 to 0.033] | 0.079 [0.062 to 0.097]
  Rectal Biopsy-Male-Visit 2: number analyzed (Participants) | 5 | 6
  Rectal Biopsy-Male-Visit 2 | 0.00095 [0.00093 to 0.00095] | 0.00092 [0.00086 to 0.0012]
  Rectal Biopsy-Male-Visit 4: number analyzed (Participants) | 5 | 7
  Rectal Biopsy-Male-Visit 4 | 0.14 [0.12 to 0.15] | 0.25 [0.18 to 0.47]
  Rectal Biopsy-Male-Visit 8: number analyzed (Participants) | 3 | 5
  Rectal Biopsy-Male-Visit 8 | 0.21 [0.17 to 0.22] | 0.6 [0.54 to 0.61]
  Rectal Biopsy-Male-Visit 9: number analyzed (Participants) | 4 | 6
  Rectal Biopsy-Male-Visit 9 | 0.027 [0.016 to 0.034] | 0.047 [0.03 to 0.078]
  Rectal Secretions-Female-Visit 2: number analyzed (Participants) | 6 | 6
  Rectal Secretions-Female-Visit 2 | 0.0024 [0.0022 to 0.0029] | 0.0026 [0.0019 to 0.0036]
  Rectal Secretions-Female-Visit 4: number analyzed (Participants) | 6 | 6
  Rectal Secretions-Female-Visit 4 | 0.0025 [0.0017 to 0.0027] | 0.003 [0.0026 to 0.0037]
  Rectal Secretions-Female-Visit 5: number analyzed (Participants) | 6 | 5
  Rectal Secretions-Female-Visit 5 | 0.002 [0.0016 to 0.0025] | 0.0024 [0.002 to 0.0048]
  Rectal Secretions-Female-Visit 6: number analyzed (Participants) | 6 | 6
  Rectal Secretions-Female-Visit 6 | 0.0039 [0.0025 to 0.0049] | 0.0035 [0.0026 to 0.0042]
  Rectal Secretions-Female-Visit 7: number analyzed (Participants) | 5 | 6
  Rectal Secretions-Female-Visit 7 | 0.0028 [0.0024 to 0.0033] | 0.0029 [0.0024 to 0.003]
  Rectal Secretions-Female-Visit 8: number analyzed (Participants) | 6 | 6
  Rectal Secretions-Female-Visit 8 | 0.0037 [0.0028 to 0.0041] | 0.0026 [0.002 to 0.0028]
  Rectal Secretions-Female-Visit 9: number analyzed (Participants) | 6 | 4
  Rectal Secretions-Female-Visit 9 | 0.0027 [0.0023 to 0.003] | 0.0031 [0.0024 to 0.0035]
  Rectal Secretions-Male-Visit 2: number analyzed (Participants) | 5 | 7
  Rectal Secretions-Male-Visit 2 | 0.0039 [0.0031 to 0.0048] | 0.003 [0.0016 to 0.0034]
  Rectal Secretions-Male-Visit 4: number analyzed (Participants) | 4 | 7
  Rectal Secretions-Male-Visit 4 | 0.0032 [0.0029 to 0.0033] | 0.0027 [0.0022 to 0.0034]
  Rectal Secretions-Male-Visit 5: number analyzed (Participants) | 4 | 6
  Rectal Secretions-Male-Visit 5 | 0.0045 [0.0036 to 0.0074] | 0.0029 [0.002 to 0.0038]
  Rectal Secretions-Male-Visit 6: number analyzed (Participants) | 4 | 6
  Rectal Secretions-Male-Visit 6 | 0.004 [0.0032 to 0.0046] | 0.0025 [0.0019 to 0.0037]
  Rectal Secretions-Male-Visit 7: number analyzed (Participants) | 4 | 6
  Rectal Secretions-Male-Visit 7 | 0.0035 [0.0031 to 0.004] | 0.0038 [0.003 to 0.0046]
  Rectal Secretions-Male-Visit 8: number analyzed (Participants) | 3 | 4
  Rectal Secretions-Male-Visit 8 | 0.004 [0.003 to 0.0043] | 0.0043 [0.0039 to 0.0048]
  Rectal Secretions-Male-Visit 9: number analyzed (Participants) | 4 | 6
  Rectal Secretions-Male-Visit 9 | 0.0032 [0.0027 to 0.0036] | 0.0034 [0.0029 to 0.0041]
  Semen-Male-Visit 2: number analyzed (Participants) | 5 | 7
  Semen-Male-Visit 2 | 0.000044 [0.000036 to 0.000044] | 0.000048 [0.000045 to 0.000053]
  Semen-Male-Visit 4: number analyzed (Participants) | 5 | 7
  Semen-Male-Visit 4 | 0.02 [0.014 to 0.02] | 0.04 [0.027 to 0.049]
  Semen-Male-Visit 5: number analyzed (Participants) | 4 | 6
  Semen-Male-Visit 5 | 0.0028 [0.0027 to 0.0043] | 0.0082 [0.0057 to 0.011]
  Semen-Male-Visit 6: number analyzed (Participants) | 4 | 6
  Semen-Male-Visit 6 | 0.025 [0.024 to 0.026] | 0.058 [0.044 to 0.076]
  Semen-Male-Visit 7: number analyzed (Participants) | 4 | 6
  Semen-Male-Visit 7 | 0.0034 [0.003 to 0.0047] | 0.0078 [0.0045 to 0.0097]
  Semen-Male-Visit 8: number analyzed (Participants) | 3 | 5
  Semen-Male-Visit 8 | 0.02 [0.017 to 0.02] | 0.056 [0.036 to 0.057]
  Semen-Male-Visit 9: number analyzed (Participants) | 4 | 6
  Semen-Male-Visit 9 | 0.005 [0.0045 to 0.0054] | 0.0091 [0.0045 to 0.015]
  Softcup Fluid-Female-Visit 2: number analyzed (Participants) | 4 | 5
  Softcup Fluid-Female-Visit 2 | 0.00043 [0.00033 to 0.0014] | 0.00025 [0.000067 to 0.0038]
  Softcup Fluid-Female-Visit 4: number analyzed (Participants) | 5 | 5
  Softcup Fluid-Female-Visit 4 | 0.16 [0.041 to 0.4] | 0.32 [0.21 to 1.58]
  Softcup Fluid-Female-Visit 5: number analyzed (Participants) | 5 | 3
  Softcup Fluid-Female-Visit 5 | 0.017 [0.01 to 0.036] | 0.051 [0.038 to 0.083]
  Softcup Fluid-Female-Visit 6: number analyzed (Participants) | 5 | 6
  Softcup Fluid-Female-Visit 6 | 0.22 [0.18 to 0.25] | 0.36 [0.21 to 0.46]
  Softcup Fluid-Female-Visit 7: number analyzed (Participants) | 5 | 4
  Softcup Fluid-Female-Visit 7 | 0.047 [0.025 to 0.077] | 0.1 [0.015 to 0.31]
  Softcup Fluid-Female-Visit 8: number analyzed (Participants) | 5 | 6
  Softcup Fluid-Female-Visit 8 | 0.18 [0.13 to 0.21] | 0.32 [0.26 to 0.91]
  Softcup Fluid-Female-Visit 9: number analyzed (Participants) | 2 | 3
  Softcup Fluid-Female-Visit 9 | 0.021 [0.014 to 0.029] | 0.011 [0.0069 to 0.028]
  Vaginal Biopsy-Female-Visit 2: number analyzed (Participants) | 6 | 6
  Vaginal Biopsy-Female-Visit 2 | 0.0016 [0.0015 to 0.0021] | 0.003 [0.0017 to 0.0038]
  Vaginal Biopsy-Female-Visit 4: number analyzed (Participants) | 6 | 4
  Vaginal Biopsy-Female-Visit 4 | 0.14 [0.1 to 0.18] | 0.34 [0.22 to 0.47]
  Vaginal Biopsy-Female-Visit 8: number analyzed (Participants) | 6 | 5
  Vaginal Biopsy-Female-Visit 8 | 0.17 [0.13 to 0.23] | 0.26 [0.0038 to 0.28]
  Vaginal Biopsy-Female-Visit 9: number analyzed (Participants) | 5 | 4
  Vaginal Biopsy-Female-Visit 9 | 0.04 [0.0036 to 0.068] | 0.036 [0.0048 to 0.071]

12. Primary Outcome: Unnormalized Levels of VRC07-523LS in Serum Out to Week 48, 16 Weeks After the Last Product Administration
Description: Pharmacokinetic - Binding Antibody Multiplex Assay (PK-BAMA) was used to measure levels of passively infused VRC07-523LS broadly neutralizing monoclonal antibody in participant sera using 5C9 anti-IDiotype antibody (anti-ID). Outcome measure is the concentration of VRC07-523LS.
Time Frame: Measured at Visits 2, 4, 5, 6, 7, 8, 9 (Weeks -2, 2, 16, 18, 32, 34, 48).
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: µg/mL
Arm/Group | Group 1: Vaccine | Group 2: Vaccine
Number analyzed (Participants) | 11 | 13
µg/mL
  Serum-Female-Visit 2: number analyzed (Participants) | 6 | 6
  Serum-Female-Visit 2 | 0.02 [0.02 to 0.02] | 0.02 [0.02 to 0.02]
  Serum-Female-Visit 4: number analyzed (Participants) | 6 | 6
  Serum-Female-Visit 4 | 100.34 [97.99 to 120.64] | 220.14 [173.90 to 254.30]
  Serum-Female-Visit 5: number analyzed (Participants) | 6 | 5
  Serum-Female-Visit 5 | 19.23 [18.59 to 19.45] | 44.32 [31.12 to 57.41]
  Serum-Female-Visit 6: number analyzed (Participants) | 6 | 6
  Serum-Female-Visit 6 | 123.43 [120.51 to 138.82] | 249.19 [245.33 to 252.01]
  Serum-Female-Visit 7: number analyzed (Participants) | 5 | 6
  Serum-Female-Visit 7 | 22.5 [20.77 to 23.50] | 30.69 [9.35 to 56.12]
  Serum-Female-Visit 8: number analyzed (Participants) | 6 | 6
  Serum-Female-Visit 8 | 135.99 [119.09 to 151.77] | 270.93 [233.77 to 325.09]
  Serum-Female-Visit 9: number analyzed (Participants) | 6 | 4
  Serum-Female-Visit 9 | 19.71 [18.36 to 21.02] | 43.74 [41.11 to 47.69]
  Serum-Male-Visit 2: number analyzed (Participants) | 5 | 7
  Serum-Male-Visit 2 | 0.02 [0.02 to 0.02] | 0.02 [0.02 to 0.02]
  Serum-Male-Visit 4: number analyzed (Participants) | 5 | 7
  Serum-Male-Visit 4 | 95.44 [73.30 to 122.31] | 271.78 [208.78 to 296.46]
  Serum-Male-Visit 5: number analyzed (Participants) | 4 | 6
  Serum-Male-Visit 5 | 16.7 [15.15 to 19.06] | 46.43 [28.02 to 51.84]
  Serum-Male-Visit 6: number analyzed (Participants) | 4 | 6
  Serum-Male-Visit 6 | 130.3 [118.59 to 141.06] | 325.21 [285.95 to 332.78]
  Serum-Male-Visit 7: number analyzed (Participants) | 4 | 6
  Serum-Male-Visit 7 | 23.9 [18.96 to 27.94] | 45.05 [24.61 to 59.00]
  Serum-Male-Visit 8: number analyzed (Participants) | 3 | 5
  Serum-Male-Visit 8 | 132.29 [121.83 to 155.23] | 338.5 [302.74 to 378.46]
  Serum-Male-Visit 9: number analyzed (Participants) | 4 | 6
  Serum-Male-Visit 9 | 25.34 [23.50 to 27.18] | 40.44 [16.55 to 63.11]

13. Primary Outcome: IgG-normalized Levels of VRC07-523LS in Serum Out to Week 48, 16 Weeks After the Last Product Administration
Description: Pharmacokinetic - Binding Antibody Multiplex Assay (PK-BAMA) was used to measure levels of passively infused VRC07-523LS broadly neutralizing monoclonal antibody in participant sera using 5C9 anti-IDiotype antibody (anti-ID). Outcome measure is the IgG-normalized VRC07-523LS levels performed by dividing VRC07-523LS levels (pg/mL) by the average reference values for total IgG concentrations in serum in the USA (11,650,000 ng/mL).
Time Frame: Measured at Visits 2, 4, 5, 6, 7, 8, 9 (Weeks -2, 2, 16, 18, 32, 34, 48).
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: pg mAb/ng total IgG
Arm/Group | Group 1: Vaccine | Group 2: Vaccine
Number analyzed (Participants) | 11 | 13
pg mAb/ng total IgG
  Serum-Female-Visit 2: number analyzed (Participants) | 6 | 6
  Serum-Female-Visit 2 | 0.002 [0.002 to 0.002] | 0.002 [0.002 to 0.002]
  Serum-Female-Visit 4: number analyzed (Participants) | 6 | 6
  Serum-Female-Visit 4 | 8.61 [8.41 to 10.36] | 18.9 [14.93 to 21.83]
  Serum-Female-Visit 5: number analyzed (Participants) | 6 | 5
  Serum-Female-Visit 5 | 1.65 [1.6 to 1.67] | 3.8 [2.67 to 4.93]
  Serum-Female-Visit 6: number analyzed (Participants) | 6 | 6
  Serum-Female-Visit 6 | 10.59 [10.34 to 11.92] | 21.39 [21.06 to 21.63]
  Serum-Female-Visit 7: number analyzed (Participants) | 5 | 6
  Serum-Female-Visit 7 | 1.93 [1.78 to 2.02] | 2.63 [0.8 to 4.82]
  Serum-Female-Visit 8: number analyzed (Participants) | 6 | 6
  Serum-Female-Visit 8 | 11.67 [10.22 to 13.03] | 23.26 [20.07 to 27.9]
  Serum-Female-Visit 9: number analyzed (Participants) | 6 | 4
  Serum-Female-Visit 9 | 1.69 [1.58 to 1.8] | 3.75 [3.53 to 4.09]
  Serum-Male-Visit 2: number analyzed (Participants) | 5 | 7
  Serum-Male-Visit 2 | 0.002 [0.002 to 0.002] | 0.002 [0.002 to 0.002]
  Serum-Male-Visit 4: number analyzed (Participants) | 5 | 7
  Serum-Male-Visit 4 | 8.19 [6.29 to 10.5] | 23.33 [17.92 to 25.45]
  Serum-Male-Visit 5: number analyzed (Participants) | 4 | 6
  Serum-Male-Visit 5 | 1.43 [1.3 to 1.64] | 3.99 [2.4 to 4.45]
  Serum-Male-Visit 6: number analyzed (Participants) | 4 | 6
  Serum-Male-Visit 6 | 11.18 [10.18 to 12.11] | 27.92 [24.55 to 28.56]
  Serum-Male-Visit 7: number analyzed (Participants) | 4 | 6
  Serum-Male-Visit 7 | 2.05 [1.63 to 2.4] | 3.87 [2.11 to 5.06]
  Serum-Male-Visit 8: number analyzed (Participants) | 3 | 5
  Serum-Male-Visit 8 | 11.36 [10.46 to 13.32] | 29.06 [25.99 to 32.49]
  Serum-Male-Visit 9: number analyzed (Participants) | 4 | 6
  Serum-Male-Visit 9 | 2.18 [2.02 to 2.33] | 3.47 [1.42 to 5.42]

14. Primary Outcome: Protein-normalized Levels of VRC07-523LS in Serum Out to Week 48, 16 Weeks After the Last Product Administration
Description: Pharmacokinetic - Binding Antibody Multiplex Assay (PK-BAMA) was used to measure levels of passively infused VRC07-523LS broadly neutralizing monoclonal antibody in participant sera using 5C9 anti-idiotype antibody (anti-ID). Outcome measure is the protein-normalized VRC07-523LS levels performed by dividing VRC07-523LS levels (pg/mL) by the total protein (ng/mL).
Time Frame: Measured at Visits 2, 4, 5, 6, 7, 8, 9 (Weeks -2, 2, 16, 18, 32, 34, 48).
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: pg mAb/ng total protein
Arm/Group | Group 1: Vaccine | Group 2: Vaccine
Number analyzed (Participants) | 11 | 13
pg mAb/ng total protein
  Serum-Female-Visit 2: number analyzed (Participants) | 6 | 6
  Serum-Female-Visit 2 | 0.00022 [0.00022 to 0.00022] | 0.00026 [0.00025 to 0.00027]
  Serum-Female-Visit 4: number analyzed (Participants) | 6 | 6
  Serum-Female-Visit 4 | 0.97 [0.92 to 1.22] | 2.32 [1.95 to 2.69]
  Serum-Female-Visit 5: number analyzed (Participants) | 6 | 5
  Serum-Female-Visit 5 | 0.19 [0.18 to 0.2] | 0.45 [0.34 to 0.58]
  Serum-Female-Visit 6: number analyzed (Participants) | 6 | 6
  Serum-Female-Visit 6 | 1.25 [1.23 to 1.37] | 2.56 [2.54 to 2.78]
  Serum-Female-Visit 7: number analyzed (Participants) | 5 | 6
  Serum-Female-Visit 7 | 0.22 [0.21 to 0.25] | 0.35 [0.1 to 0.56]
  Serum-Female-Visit 8: number analyzed (Participants) | 6 | 6
  Serum-Female-Visit 8 | 1.3 [1.13 to 1.49] | 3 [2.81 to 3.47]
  Serum-Female-Visit 9: number analyzed (Participants) | 6 | 4
  Serum-Female-Visit 9 | 0.2 [0.19 to 0.21] | 0.49 [0.45 to 0.56]
  Serum-Male-Visit 2: number analyzed (Participants) | 5 | 7
  Serum-Male-Visit 2 | 0.00025 [0.00025 to 0.00026] | 0.00023 [0.00023 to 0.00025]
  Serum-Male-Visit 4: number analyzed (Participants) | 5 | 7
  Serum-Male-Visit 4 | 1 [0.78 to 1.33] | 2.74 [2.17 to 2.98]
  Serum-Male-Visit 5: number analyzed (Participants) | 4 | 6
  Serum-Male-Visit 5 | 0.19 [0.17 to 0.2] | 0.49 [0.31 to 0.59]
  Serum-Male-Visit 6: number analyzed (Participants) | 4 | 6
  Serum-Male-Visit 6 | 1.33 [1.22 to 1.41] | 3.08 [2.89 to 3.71]
  Serum-Male-Visit 7: number analyzed (Participants) | 4 | 6
  Serum-Male-Visit 7 | 0.24 [0.19 to 0.28] | 0.45 [0.22 to 0.58]
  Serum-Male-Visit 8: number analyzed (Participants) | 3 | 5
  Serum-Male-Visit 8 | 1.46 [1.29 to 1.63] | 3.08 [3.05 to 3.86]
  Serum-Male-Visit 9: number analyzed (Participants) | 4 | 6
  Serum-Male-Visit 9 | 0.25 [0.23 to 0.27] | 0.35 [0.16 to 0.54]

15. Secondary Outcome: Serum Concentration of ADA in Each Group Measured at Multiple Timepoints From Baseline Through the Final Study Visit
Description: Anti-drug dependent antibodies were measured by an ADA assay from specimens obtained from all participants. Tier 3 titers are only available for those participants who had positive for ADA Tiers 1 and 2.
Time Frame: Measured at Visits 2, 3, 5, 7, and 9 (Weeks -2, 0, 16, 32, 48). However, Tier 3 ADA titers are only assessed and reported at Visits 2 and 3 (Weeks -2 and 0) for the subset of participants who tested positive for ADA Tiers 1 and 2.
Population: Overall Number of Participants Analyzed represents the total number of infused participants in each group. Number Analyzed-shows the number of participants with available data after filtering for assay specific quality control criteria at each timepoint.
Measure: Median (Inter-Quartile Range); unit: Titer
Arm/Group | Group 1: Vaccine | Group 2: Vaccine
Number analyzed (Participants) | 11 | 13
Titer
  VRC07-523LS-Tier 3-Visit 2: number analyzed (Participants) | 2 | 2
  VRC07-523LS-Tier 3-Visit 2 | 15 [9.00 to 21.00] | 54 [40.50 to 67.50]
  VRC07-523LS-Tier 3-Visit 3: number analyzed (Participants) | 2 | 1
  VRC07-523LS-Tier 3-Visit 3 | 15 [9.00 to 21.00] | 27 [27.00 to 27.00]

ADVERSE EVENTS:
Time Frame: Enrollment through week 48
Description: Number of Participants Reporting Adverse Events (AEs)
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Pre-treatment
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/13 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/13 | 0/4
Other Adverse Events (participants affected / at risk) | 10/11 | 12/13 | 0/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Vaccine (N=11) | Group 2: Vaccine (N=13) | Group 3: Pre-treatment (N=4)
Any Event in SOC (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Any Event in SOC (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Chalazion (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Any Event in SOC (Gastrointestinal disorders) | 4 (4) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oral pruritus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Any Event in SOC (General disorders) | 2 (2) | 1 (1) | 0 (0)
Feeling cold (General disorders) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 1 (1) | 0 (0)
Any Event in SOC (Infections and infestations) | 9 (24) | 5 (5) | 0 (0)
Bacterial vaginosis (Infections and infestations) | 3 (4) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Molluscum contagiosum (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 8 (11) | 3 (3) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 2 (4) | 0 (0) | 0 (0)
Any Event in SOC (Injury, poisoning and procedural complications) | 3 (4) | 7 (7) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (3) | 5 (5) | 0 (0)
Muscle injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Post procedural swelling (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Any Event in SOC (Investigations) | 3 (6) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Smear cervix abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Any Event in SOC (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Any Event in SOC (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Coccydynia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Any Event in SOC (Nervous system disorders) | 3 (3) | 4 (4) | 0 (0)
Disturbance in attention (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness postural (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Any Event in SOC (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Any Event in SOC (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Any Event in SOC (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Any Event in SOC (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (4):
  • Study Protocol (2018-09-18): https://cdn.clinicaltrials.gov/large-docs/49/NCT03735849/Prot_001.pdf
  • Statistical Analysis Plan: Safety (2021-08-16): https://cdn.clinicaltrials.gov/large-docs/49/NCT03735849/SAP_002.pdf
  • Statistical Analysis Plan: Pharmacokinetics (2025-02-19): https://cdn.clinicaltrials.gov/large-docs/49/NCT03735849/SAP_003.pdf
  • Informed Consent Form (2018-09-18): https://cdn.clinicaltrials.gov/large-docs/49/NCT03735849/ICF_000.pdf